CLINICAL TRIAL: NCT04867421
Title: Assessment of the Presence, and Characterization, of Tumor-associated Neutrophils in Bone Sarcomas: Pilot Study
Brief Title: Neutrophils in Bone Sarcomas
Acronym: TANOs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-003-TANOs
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Osteosarcoma, Chondrosarcoma
Keywords: Osteosarcoma; Chondrosarcoma; Tumor associated neutrophils
MeSH Terms: conditions — Osteosarcoma; Chondrosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TANOs: Adult patients with osteosarcoma or chondrosarcoma
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Hypothesis: Tumor infiltrating neutrophils are present in osteosarcomas and chondrosarcomas and

Experimental design: Exploratory observational research

Population: Adult patients with osteosarcoma or chondrosarcoma

Assessment criteria: Determination of the presence of TANs within tumors and their N1 or N2 profile, the presence of other immune cells, and the PDL-1 status of the tumor.

Investigation plan: Proposal to participate at all eligible patient during the preoperative consultation. If the patient agrees to participate in the study he/she will be included. Participation in the study will not affect its coverage. Patient participation will lead to:

* Taking samples from an operative part,
* The collection of demographic data (age, sex, height, weight, body mass index), family history of cancer, history of bone trauma, sports practice, clinical and anatomopathology reports and data, medical history (Diabetes, Cardiovascular Diseases, Infectious Diseases, Autoimmune Diseases, Bone Metabolism Disorders, Allergies, Menopause, Drug treatments followed, Psychiatric disorders).

Statistical analysis plan: Description in frequency of the presence of TANs, of N1 and N2 profiles, of the presence of other immune cells both qualitatively and quantitatively. Analysis in subgroups on relevant criteria (age, sex, location, type of tumor).

ELIGIBILITY:
Inclusion Criteria:

* Patient of 18 years and more
* Patient of the Orthopedic and Traumatological Surgery Department of the Reims University Hospital or the Godinot Institute
* Patient with osteosarcoma or chondrosarcoma to be operated on regardless of stage.
* Patient agreeing to participate in the study (informed consent form)
* Patient fluent in French
* Patient affiliated with a social security regimen

Exclusion Criteria:

* Patient having a medical history that may compromise the protocol (psychiatric, medical or pharmacological disorders such as the use of anti-inflammatory drugs, or any compound that may alter or modify the inflammatory reaction in the week preceding the protocol).
* Pregnant or breastfeeding women
* Patient with eating disorders (anorexia, bulimia, overeating)
* Patient protected by law (guardianship, curatorship, hospitalized without their consent and not protected by law, deprived of liberty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with osteosarcoma or chondrosarcoma consulting the Orthopedic and Traumatological Surgery Department of the Reims University Hospital or the Godinot Institute and undergoing tumor resection surgery
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the presence of neutrophils in sarcoma-affected tissues | Time of surgery
  Flow cytometry analysis on excised tissues

SECONDARY OUTCOMES:
Comparison of flow cytometry and histology for neutrophil assessment in sarcoma-affected tissues | Time of surgery
  Neutrophil identification thanks to CD66b marker with both the techniques
Identification of neutrophils N1 or N2 profile in sarcoma-affected tissues | Time of surgery
  Flow cytometry (CD45 CD66b CD182 CD184 CD195)
Identification of non-neutrophil leukocytes in sarcoma-affected tissues | Time of surgery
  Flow cytometry analysis (CD45 CD3 CD4 CD8 CD19 CD33 CD80 CD163)
Determination of PDL1 status of neutrophils in sarcoma-affected tissues | Time of surgery
  Flow cytometry analysis (CD45 CD66b CD 274)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe MESA, Principal Investigator — Université de Reims Champagne-Ardenne - CHU de Reims
Locations (1):
- Université de Reims Champagne-Ardenne, Reims, France